CLINICAL TRIAL: NCT02881502
Title: Clinical Study of Relationship Between Granulocyte Activation, HDAC2 and Severe Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Haiqin Guo, Master Degree Candidate,Student of Respiratory Medicine, Xijing Hospital
Other Study IDs: Haiqin Guo
Record Dates: First submitted 2016-07-15; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: granulocyte activation; HDAC2; severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy control group: Mainly from students, family members of patients without chronic lung disease, healthy population, age 18-75 years old, the gender is not limited.
- mild and moderate asthma group: Patients diagnosed with asthma in the outpatient clinic, in accordance with the inclusion criteria and exclusion criteria.
- severe asthma group: Outpatient patients with severe asthma diagnosis, in accordance with the inclusion criteria and exclusion criteria.
  Interventions: Other: severe asthma group

INTERVENTIONS:
Other: severe asthma group — No intervention
  Groups: severe asthma group

SUMMARY:
Program： Clinical Study of Relationship Between Granulocyte Activation, HDAC2 and Severe Asthma Aim：The early prediction of severe asthma, early intervention on the disease, reduce the family and the national finance.

design:This study is a single center randomized controlled trial designed by the Department of respiratory medicine, Xijing Hospital, as the main research unit.Compare the case group(severe asthma group and mild-and-moderate asthma group) and control group(healthy control group) by detecting the activity of MPO、NE、MMP-9 and ECP in the peripheral blood and the activity of HDAC2 in PBMCs of patients.

case:60

Case selection:

Inclusion criteria: age 18-75 years old; diagnosis of asthma was clear; informed consent was signed.

Exclusion criteria: poor compliance; cognitive ability is low; psychiatric disorders need to be combined with psychotropic medication.

DETAILED DESCRIPTION:
Application of SPSS 19 statistical software. Measurement data were expressed as mean ± standard deviation.

First the data is normality tested and homogeneity of variance tested, according to the measurement data of normal distribution by SNK single factor analysis of variance; does not conform to the normal distribution of measurement data, using the Kruskal Wallis non parametric test. P < 0.05 for the difference was statistically significant.

ELIGIBILITY:
inclusion criteria: healthy control group：

* Mainly from students,
* family members of patients without chronic lung disease,
* healthy population,
* age 18-75 years old, the gender is not limited. case group：
* The patient has been diagnosed with asthma in the outpatient clinic. The diagnostic criteria are in accordance with the Guidelines for Prevention and Treatment of Bronchial Asthma in the respiratory disease branch of the Chinese Medical Association.

In the past 1 year need guidelines of global asthma record instrument 4-5 drug treatment of asthma [high dose inhaled corticosteroid with long-acting beta2 receptor agonist or leukotriene modifiers / theophylline or systemic hormone therapy is more than or equal to 50% of the time, in order to prevent into uncontrolled asthma, or even in the treatment is to control asthma patients for severe asthma.

exclusion criteria：

* Poor treatment compliance, or low cognitive ability to impact the self rating scale ;
* There are serious heart, liver, renal dysfunction, or other infectious diseases ;
* The individual who refuse to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatients and the students
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite severe asthma confirmed by the plasma concentration of blood related indexes(MPO、MMP-9、NE、ECP、HDAC2) | one year
  Compare the difference was not statistically significant of the different groups by testing the concentration of blood related indicators of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Wu C gui, professor, Study Director — Xijing Hospital
Locations (1):
- XijingH, Xian, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided